CLINICAL TRIAL: NCT03359954
Title: PRECISE: Preoperative Radiotherapy to Elicit Critical Immune Stimulating Effects
Brief Title: Radiation Therapy Before Surgery in Treating Patients With Hormone Receptor Positive, HER2 Negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0362; NCI-2018-00993 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0362 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-11-28; First posted 2017-12-02 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Estrogen Receptor Positive; HER2/Neu Negative; Invasive Breast Carcinoma; Progesterone Receptor Positive
MeSH Terms: interventions — Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (radiation therapy, surgery) (Experimental): Patients undergo boost radiation therapy 6-8 days before breast surgery. After surgery, patients continue to receive standard of care radiation therapy.
  Interventions: Radiation: Radiation Therapy; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; RADIOTHERAPY; RT; Therapy, Radiation
Procedure: Therapeutic Conventional Surgery — Undergo breast surgery

SUMMARY:
This phase II trial studies how well radiation therapy before surgery works in treating patients with hormone receptor positive, HER2 negative breast cancer. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the change in percent tumor-infiltrating lymphocytes (TIL) as a continuous variable before and after preoperative boost radiotherapy (RT) in hormone receptor (HR)+/human epidermal growth factor receptor2 (HER2)- breast cancers.

SECONDARY OBJECTIVES:

I. To evaluate the safety of preoperative boost RT administered to patients with HR+/HER2- breast cancer.

EXPLORATORY OBJECTIVES:

* I. To assess the mechanisms of cell death induced by preoperative boost RT.
* II. To assess immunologic and molecular responses to preoperative boost RT.
* III. To assess the correlations between immune markers, cell death markers, and their changes during treatment.
* IV. To determine if magnetic resonance imaging (MRI) can be used to predict breast tumor response to neoadjuvant radiation.

OUTLINE:

Patients undergo boost radiation therapy 6-8 days before breast surgery. After surgery, patients continue to receive standard of care radiation therapy.

After completion of study treatment, patients are followed up at 6 months.

ELIGIBILITY:
Inclusion Criteria:

Inclusion:

* Age >/=18 years at time of study entry
* Histologically confirmed HR+/HER2- (according to American Society of Clinical Oncology/College of American Pathologists guidelines) invasive carcinoma of the breast
* Presence of a clip in the primary breast cancer
* Biopsy-amenable residual disease in the breast measuring >/= 1cm in at least one dimension on ultrasound cm in at least one dimension on ultrasound
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Signed written informed consent
* Planned for multidisciplinary evaluation by a Breast Surgical Oncologist and Breast Radiation Oncologist. For patients undergoing mastectomy and desirous of reconstruction or those undergoing breast conservation in whom oncoplastic local tissue rearrangement or reduction mammoplasty is being considered, this multidisciplinary evaluation will also include a plastic surgeon.

Exclusion:

* Women who are pregnant or breast-feeding
* Contraindication to receive radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Change in Percent of Tumor-Infiltrating Lymphocytes (TIL) | 6 to 8 days after preoperative radiotherapy
  With 20 patients, a 95% confidence interval for the mean difference between TIL measurements would extend 0.44*s units from the mean (where "s" is the standard deviation of the TIL differences). If the differences are not normally distributed, researchers will report the median difference along with appropriate 95% confidence intervals. Appropriate graphs used to visualize the data.

SECONDARY OUTCOMES:
Delay Rate of Surgery Following Boost RT | 4 weeks after boost RT
  Delay rate defined as the proportion of patients experiencing a > 4 week interval between boost RT and surgery.
  The method of Thall, Simon, and Estey employed to perform interim delay rate monitoring.
Tumor Changes between pre and post boost | Up to 4 weeks after surgery
  For tumor measures, descriptive statistics including plots, tabulations, mean, median, and standard deviations will be used to summarize data. Differences and/or percentage changes will be calculated between pre- and post- therapy samples from each patient and described as continuous measures by using paired t-tests will be explored to evaluate the changes in markers pre- and post-boost therapy. Scatter plots will be used to visualize how correlated between changes in immune markers and extent of tumor cell apoptosis, and the Spearman correlation coefficients will be calculated to evaluate the association between changes in immune markers and extent of tumor cell death markers.
Toxicity calculated using the CTCAE v4.0 | 6 months after adjuvant RT
  Toxicity and cosmesis will be calculated and reported, to enable comparisons to other published reports of breast cancer-related toxicity using the CTCAE v4.0.
Changes in dynamic contrast enhanced (DCE) | 4 weeks after surgery
  Changes in DCE, internal texture, ADC values, z-spectrum asymmetry on CEST measures will be assessed between the simulation MRI and the MRI obtained following radiation boost.

CONTACTS AND LOCATIONS:
Overall Officials: Simona F Shaitelman, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org